CLINICAL TRIAL: NCT05581784
Title: The Effectiveness of a Pain Neuroscience Education Program Compared to Conventional Treatment on Pain, Biopsychosocial Variables, and Functional Capacity in Adults With Cancer Pain
Brief Title: Effectiveness of a Pain Neuroscience Education Program in Adults With Cancer Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Neurociencia Del Dolor (Other)
Collaborators: Universidad Santiago de Cali (Other); Clinica de Occidente (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INeurocienciaDolor02
Record Dates: First submitted 2022-10-01; First posted 2022-10-17 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Cancer Pain
Keywords: Pain Neuroscience education; Cancer pain; Paliative therapy; Neoplasm
MeSH Terms: conditions — Cancer Pain; Neoplasms

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Masking: Simple (result evaluator)
Who Masked: Investigator, Outcomes Assessor
Masking Description: Simple (result evaluator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain neuroscience education. (Experimental): This consists of generating elements from neurobiology and neurophysiology for the understanding of pain from the development of metaphors.
  Interventions: Other: Pain neuroscience education
- Conventional treatment or Usual Care (Other): Pharmacological treatment and indications estimated by a specialist in palliative care and pain.
  Interventions: Other: Conventional management or Usual care

INTERVENTIONS:
Other: Pain neuroscience education — PNE sessions will be led by an experienced physical therapist certified in PNE in 35-minute face-to-face group sessions. Here elements of the neurophysiology of pain are addressed, as well as the different psychosocial dimensions that influence it. The distribution of themes will be carried out as follows:
  Week One: Coping with Pain. Week 2: Pain and Cognition Week 3: Your security system Week 4: Altered Alarm System (extra sensitive). Week 5: The defense system is in distress. Week 6: Fatigue, anxiety, and stress Week 7: Current Models of Treatment Week 8: Achievements and goals Week 9: Pain emphasis and differentiation This group remains with pharmacological treatment and the usual guidelines given by the doctor.
  Other Names: Explaining Pain; Therapeutic Neuroscience Education
  Arms: Pain neuroscience education.
Other: Conventional management or Usual care — This group will only have pharmacological treatment and the usual guidelines given by the doctor. Without educational intervention.
  Other Names: Usual care; Conventional management
  Arms: Conventional treatment or Usual Care

SUMMARY:
IASP defines "pain" as "an unpleasant sensory and emotional experience associated with or resembling that associated with actual or potential tissue damage". In some patients, pain is one of the reasons they initially consult a doctor and will be strongly related to cancer itself, is connected to receiving the cancer diagnosis, and therefore may become an uncertain threat of disease recurrence in cancer survivors. Neuropathic pain is the most prevalent type of pain, but a mixed type of pain is also common, reflecting the complexity of the pain experience. There is increasing evidence in oncology that quality of life and survival are linked to early and effective palliative care, including pain management. Although improvements have been seen, undertreatment of pain remains a problem in a significant subset of cancer patients. Regarding the interventional options in cancer pain, multiple possibilities range from pharmacological modulation, the use of modalities or physical means, as well as the practice of physical exercise as a mechanism of pain modulation, which has been established according to the background grade of recommendation. Regarding education in neuroscience, this has gained momentum in chronic pain since previous interventions have generated recommendations to include neurocognitive interventions in pain processes. Therefore, it seeks to determine the effectiveness of a neuroscience education program compared to conventional treatment in adults with cancer pain in biopsychosocial variables.

DETAILED DESCRIPTION:
A parallel group randomized controlled clinical trial will be conducted during the months of November 2022 to December 2023. The proposed research will be a quantitative experimental design type controlled clinical trial following the SPIRIT guidelines for clinical trial protocols and CONSORT for the execution of clinical trials.

A total of 80 patients, where 40 will be assigned to (PNE) and 40 to conventional management. experimental group: based on education in neuroscience of pain for 9 sessions in a period of 10 weeks. Work will be done to prepare the content for an adapted and illustrated guide as a complementary material for patients. An expert judgment test will be carried out to validate the content of the material. Each patient must complete at least 8 sessions to comply with the protocol. These sessions will be personalized and will include the guide as complementary material for each session. This group remains with pharmacological treatment and the usual guidelines given by the doctor. Results will be assessed at baseline (t1) and at week 10 (t2). Written informed consent will be obtained from all participants prior to their participation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a life expectancy of more than three months (Karnofski Scales (KPS), Eastern Cooperative Oncology Group Scale (ECOG), survival prognosis PAP score, Palliative Prognosis Index PPI).
* Acceptance of informed consent.
* Educational level (high school diploma).
* No pain hospitalizations in the previous month
* Capable of establishing a team communication process
* at least 21 points on the MOCA scale for preserved cognitive function
* Understanding of the Spanish language.

Exclusion Criteria:

* Surgery scheduled within the next three months
* Visual and auditory sensory system deficiency (deafness or blindness).
* The presence of a recent traumatic injury
* Atrial or ventricular arrhythmias that are uncontrolled.
* Aortic aneurysm dissection
* Aortic stenosis severe
* Endocarditis or pericarditis that is acute
* Uncontrollable hypertension
* Thromboembolic disease, acute.
* Acute severe heart failure
* Acute severe respiratory failure
* Fracture within the last month

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2023-12-22 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in Brief Pain Inventory (Impact of pain) | At baseline and through intervention's completion, 10 weeks
  The BPI or brief pain questionnaire is a self-administered questionnaire that contains two dimensions: one related to the intensity of pain and the impact of pain on the activities of the patient's life. Its use has increased in the evaluation of patients with cancer pain. The patient is asked to rate their worst, least, average, and current pain intensity, list current treatments and their perceived effectiveness, and rate the degree that pain interferes with general activity, mood, walking ability, normal work, relations with other persons, sleep, and enjoyment of life on a 10 point scale. the higher the score, the greater the severity of the pain.
Change in Visual Analog Scale-Pain (EVA) | At baseline and through intervention's completion, 10 weeks
  The severity of the pain at rest was assessed on a 10 cm visual analog scale (Total score: 0-10)(0=no pain, 10=severe pain) Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Change in Central Sensitization Inventory Score (CSI) | At baseline and through intervention's completion, 10 weeks
  Central Sensitization Inventory (CSI) is a scale used to detect patients with symptoms associated with central sensitization or types of central sensitization syndrome such as fibromyalgia, temporomandibular joint disease, tension type headache, migraine.
  The Central Sensitization Inventory (CSI) consists of two parts:
  Part A consists of 25 questions about central sensitization syndrome (CNS) symptoms; Section B examines the patient's condition of being diagnosed with certain CNS diseases or CNS related diseases such as anxiety and depression.
  The patient answers 25 questions in section A with a score between 0 and 4. The total score will be between 0-100. Results above 40 points indicate central sensitization.
Change in Pain Catastrophizing Scale (PCS) | At baseline and through intervention's completion, 10 weeks
  The PCS is measured with a self-administered questionnaire. Is a 13-item inventory that measures 3 elements of the perception of the intensity of pain (rumination, magnification, feeling helpless). Participants indicate the degree to which they agree with statements related their pain by selecting 0 = not at all, 1 = to a slight degree, 2 = to a moderate degree, 3 = to a great degree, 4 = all the time. There are three subscale scores assessing rumination, magnification and helplessness. All subscales are summed to produce a total score ranging from 0 to 52 with higher scores indicating the participant is having more thoughts about the pain they feel helplessness. All subscales are summed to produce a total score ranging from 0 to 52 with higher scores indicating the participant is having more thoughts about the pain they feel.
Change in Tampa Scale for Kinesiophobia (TSK-11) | At baseline and through intervention's completion, 10 weeks
  TSK-11 is used to assess fear of pain and movement. It consists of 11 items, which are answered on a Likert scale of 4 points. Total scores of each scale range from 11 to 44, where higher scores indicate a greater fear of pain and movement.
Change in Beck Depression Inventory Score | At baseline and through intervention's completion, 10 weeks
  Beck Depression Criterion (BDI) is a commonly used evaluation criterion for diagnosis and follow-up parameters in assessing depression status.It contains 21 categories to measure physical, emotional, cognitive and motivational symptoms such as hopelessness, irritability, guilt, feeling of punishment, fatigue, and weight loss in each depression, and each category is scored between 0-3. The patient is asked to mark the most appropriate one for the four options in each category. Scoring progressively increases from the absence of symptoms to severe symptoms. 0-10 points: No depression, 11-17 points: Mild depression, 18-23 points: Moderate depression, 24 and above points: Severe depression.
Change in DN4 neuropathic pain | At baseline and through intervention's completion, 10 weeks
  We will work with the DN4 scale that evaluates 4 questions with a possibility of being qualified up to 10 points to determine the presence of neuropathic pain.
Change in Moca test Cognitive function | At baseline and through intervention's completion, 10 weeks
  It is made up of 19 items and eight cognitive domains that assess skills such as visuospatial/executive, naming, memory, attention, language, abstraction, delayed recall, and orientation. a maximum score of 30, with the cut-off points for cognitive impairment being 25/26.
Change in EORTC QLQ C-30 Quality of life | At baseline and through intervention's completion, 10 weeks
  has been defined as the way in which the individual perceives his/her place in life, The standard model consists of 14 domains and an empirical solution with five domains (physical, psychological, frailty, socioeconomic, and global score). This widely used questionnaire consists of five functional scales (physical, role, cognitive, emotional, and social function), a global quality of life (QoL) scale, three symptom scales (fatigue, nausea and vomiting, and pain), and six individual. items (loss of appetite, diarrhea, dyspnea, constipation, insomnia, economic impact). For the functional and global quality of life scales, a higher score indicates better health. For the symptom scales, a higher score indicates a higher symptom burden.
Change in Sleep quality Pittsburgh Sleep Quality Index | At baseline and through intervention's completion, 10 weeks
  This is one of the most reliable tests to define the quality of sleep and its disorders. It contains a total of 19 questions, grouped into 10 questions. The questions are combined to form seven areas with their corresponding score, each one of which shows a range between 0 and 3 points.

OTHER OUTCOMES:
Change in 6-minute walk test | At baseline and through intervention's completion, 10 weeks
  It is performed to determine exercise tolerance and specify functional status. This evaluates the number of meters traveled during the last 6 minutes.
Change in grip strength | At baseline and through intervention's completion, 10 weeks
  It is a marker of nutritional status and a marker of morbidity and mortality of the pathology. It will be measured with a dynamometer to establish the grip strength value in kilograms.
Change in Test Get up and Go | At baseline and through intervention's completion, 10 weeks
  This test has been developed, finding that it has been a predictor of falls and as a measure of functional capacity. n this test, the participant starts in a chair, stands up, runs three meters, and sits down again. The time of the execution of the test is taken.

CONTACTS AND LOCATIONS:
Locations (4):
- Universidad Arturo Prat, Iquique, Chile
- Colombia (2):
  - Universidad Santiago de Cali, Cali, Valle del Cauca Department
  - Clinica de Occidente, Cali, Valle del Cauca Department
- Instituto Neurociencia del Dolor, Puebla City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nijs J, Wijma AJ, Leysen L, Pas R, Willaert W, Hoelen W, Ickmans K, Wilgen CPV. Explaining pain following cancer: a practical guide for clinicians. Braz J Phys Ther. 2019 Sep-Oct;23(5):367-377. doi: 10.1016/j.bjpt.2018.12.003. Epub 2018 Dec 21. PMID 30606621
- [Background] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884
- [Background] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c869. doi: 10.1136/bmj.c869. No abstract available. PMID 20332511
- [Derived] Ordonez-Mora LT, Rosero ID, Morales-Osorio MA, Guil R, Quintero Jordan G, Agudelo Jimenez JA, Gonzalez-Ruiz K, Avila-Valencia JC. NEUROCANTRIAL: study protocol for a randomised controlled trial of a pain neuroscience education programme in adults with cancer pain. BMJ Open. 2023 Sep 27;13(9):e071493. doi: 10.1136/bmjopen-2022-071493. PMID 37758676
- See also: Pain definition — https://www.iasp-pain.org/